CLINICAL TRIAL: NCT02045836
Title: Immunogenicity and Safety Study of GSK Biologicals' Herpes Zoster Vaccine GSK1437173A When Co-administered With Pneumovax 23™ in Adults Aged 50 Years and Older
Brief Title: Study to Evaluate Immunogenicity and Safety Study of GSK Biologicals' Herpes Zoster (HZ) Vaccine GSK1437173A When Co-administered With Pneumovax 23™ in Adults Aged 50 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 116889; 2012-005314-19 (EudraCT Number)
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Results first posted 2017-07-05 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Herpes Zoster; Herpes Zoster Vaccine
Keywords: Pneumovax 23; Co-administration; Herpes zoster; Immunogenicity; Safety; Adults
MeSH Terms: conditions — Herpes Zoster | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

ARMS (2):
- Co-Ad Group (Experimental): Subjects received one dose of the GSK1437173A study vaccine and one dose of the Pneumovax™ 23 vaccine at Day 0 and a second dose of GSK1437173A study vaccine at Month 2. GSK1437173A vaccine was administered intramuscularly, in the deltoid region of the non-dominant arm. Pneumovax™ 23 was administered intramuscularly, in the deltoid region of the dominant arm.
  Interventions: Biological: Herpes Zoster vaccine GSK 1437173A; Biological: Licensed pneumococcal polysaccharide conjugate vaccine (23-valent, adsorbed), Pneumovax 23™
- Control Group (Active Comparator): Subjects received one dose of the Pneumovax™ 23 vaccine at Day 0, one dose of the GSK1437173A study vaccine at Month 2 and a second dose of the GSK1437173A study vaccine at Month 4. GSK1437173A vaccine was administered intramuscularly, in the deltoid region of the non-dominant arm. Pneumovax™ 23 was administered intramuscularly, in the deltoid region of the dominant arm.
  Interventions: Biological: Herpes Zoster vaccine GSK 1437173A; Biological: Licensed pneumococcal polysaccharide conjugate vaccine (23-valent, adsorbed), Pneumovax 23™

INTERVENTIONS:
Biological: Herpes Zoster vaccine GSK 1437173A — 2 doses administered intramuscularly (IM) in the deltoid region of the non-dominant arm.
Biological: Licensed pneumococcal polysaccharide conjugate vaccine (23-valent, adsorbed), Pneumovax 23™ — One dose administered intramuscularly (IM) in the deltoid region of the non-dominant arm.
  Other Names: Pneumo 23™

SUMMARY:
The purpose of this study is to assess the immunogenicity, reactogenicity and safety of the GSK Biologicals HZ/su candidate vaccine when its first dose is co-administered with Pneumovax 23™ vaccine in adults aged 50 years or older.The impact of HZ/su vaccine on Pneumovax 23™ vaccine immune response will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female aged 50 years or older at the time of the first vaccination with the study vaccine(s).
* Written informed consent obtained from the subject.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. A prednisone dose of < 20 mg/day is allowed. Inhaled, topical and intra-articular corticosteroids are allowed.
* Administration or planned administration of a vaccine not foreseen by the study protocol within the period starting 30 days before the first dose of study vaccine(s) and ending 30 days after the last dose of study vaccine. This includes any type of vaccine such as live, inactivated and subunit vaccines.
* Administration of long-acting immune-modifying drugs within six months prior to the first vaccine dose or expected administration at any time during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Previous vaccination against Varicella-zoster virus (VZV) or HZ and/or planned administration during the study of an HZ or VZV vaccine other than the study vaccine.
* History of HZ.
* History of documented pneumococcal infection within 5 previous years.
* Prior receipt of any pneumococcal vaccine or planned use of this vaccine during the study period, other than the study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy .
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 37.5°C /99.5°F by oral route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions before 2 months after the last dose of study vaccine.
* Any persons with cerebrospinal fluid (CSF) leaks, cochlear implants, chronic renal failure, nephrotic syndrome, and functional or anatomic asplenia.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.
* Any condition which, in the judgment of the investigator, would make intramuscular (IM) injection unsafe.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 865 (Actual)
Dates: Start 2014-03-05 (Actual); Primary Completion 2015-07-02 (Actual); Study Completion 2016-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (3):
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Columbia, Maryland
- Canada (3):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu

REFERENCES:
- [Background] Marechal C, Lal H, Poder A, Ferguson M, Enweonye I, Heineman TC, Herve C, Rheault P, Talli J, Wauters D, Oostvogels L. Immunogenicity and safety of the adjuvanted recombinant zoster vaccine co-administered with the 23-valent pneumococcal polysaccharide vaccine in adults >/=50 years of age: A randomized trial. Vaccine. 2018 Jul 5;36(29):4278-4286. doi: 10.1016/j.vaccine.2018.05.110. Epub 2018 Jun 11. PMID 29903674

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Co-Ad Group | Control Group
Started | 432 | 433
Completed | 423 | 419
Not Completed | 9 | 14
Not completed — Adverse Event | 4 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 4 | 7
Not completed — Migrated from study area | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Co-Ad Group | Control Group | Total
Number analyzed (Participants) | 432 | 433 | 865
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (8.4) | 63.2 (8.4) | 63.2 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 264 | 252 | 516
  Male | 168 | 181 | 349
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian / European Heritage | 408 | 406 | 814
  African Heritage / African American | 12 | 9 | 21
  American Indian or Alaskan Native | 1 | 3 | 4
  Asian - East Asian Heritage | 3 | 7 | 10
  Asian - Japanese Heritage | 0 | 1 | 1
  Asian - South East Asian Heritage | 4 | 2 | 6
  White - Arabic / North African Heritage | 2 | 0 | 2
  Mixed Origin | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Vaccine Response for Anti-gE Antibodies
Description: Vaccine response rate for anti-gE antibody concentrations, as determined by enzyme-linked immunosorbent assay (ELISA), in subjects from the Co-Ad group. Vaccine response defined as : For initially seronegative subjects, antibody concentration at post-vaccination ≥ 4 fold the cut-off for Anti-gE (4x97 mIU/mL) For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4 fold the pre-vaccination antibody concentration
Time Frame: At Month 3
Population: This analysis was perfrmed on the According-to-Protocol (ATP) cohort for immunigenicity, which included all evaluable subjects who met all eligibility criteria, who complied with the procedures and intervals allowed for the analysis, not eliminated during the study and for whom data concerning immunogenicity endpoint measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group
Number analyzed (Participants) | 401
Participants | 394

2. Primary Outcome: Anti-glicoprotein E (gE) Antibody Concentrations
Description: Antibody concentrations were determined by ELISA, presented as geometric mean concentrations and expressed as milli international units per milliliter (mIU/mL).
Time Frame: At one month post-dose 2 (Month 3 for the Co-Ad Group and Month 5 for the Control Group)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 407 | 402
mIU/mL | 49918.0 [47143.0 to 52856.3] | 50327.9 [47200.4 to 53662.7]

3. Primary Outcome: Anti-pneumococcal Antibody Titers
Description: Anti-pneumococcal antibody titers were presented as geometric mean titers (GMTs) for the 12 following serotypes as determined by Opsonophagocytic Assay (OPA): 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F.
Time Frame: At one month post-dose (Month 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 410 | 413
Titers
  MOPA-1 | 65.1 [54.2 to 78.1] | 68.6 [56.9 to 82.7]
  MOPA-9V | 1898.4 [1618.1 to 2227.2] | 1991.3 [1716.0 to 2310.8]
  MOPA-14 | 2629.4 [2297.4 to 3009.3] | 2612.8 [2230.7 to 3060.3]
  MOPA-3 | 106.7 [92.6 to 122.9] | 107.4 [92.7 to 124.4]
  MOPA-4: number analyzed (Participants) | 410 | 412
  MOPA-4 | 1079.4 [924.0 to 1260.9] | 1328.8 [1141.0 to 1547.6]
  MOPA-5 | 161.4 [134.6 to 193.6] | 149.5 [123.5 to 181.0]
  MOPA-6B | 1619.0 [1354.5 to 1935.0] | 1564.4 [1303.5 to 1877.6]
  MOPA-7F | 2352.5 [2049.5 to 2700.3] | 2460.4 [2128.7 to 2843.8]
  MOPA-18C: number analyzed (Participants) | 409 | 413
  MOPA-18C | 1077.4 [921.1 to 1260.2] | 1076.0 [918.2 to 1260.9]
  MOPA-19A: number analyzed (Participants) | 409 | 413
  MOPA-19A | 1349.6 [1152.1 to 1580.8] | 1573.1 [1350.7 to 1832.2]
  MOPA-19F | 904.3 [779.6 to 1049.0] | 953.0 [814.8 to 1114.6]
  MOPA-23F | 431.4 [356.1 to 522.7] | 367.3 [300.8 to 448.5]

4. Primary Outcome: Adjusted Ratios of Geometric Mean Titers (GMTs) Between Groups
Description: The Adjusted ratios of GMTs between groups (Control group and Co-Ad group) were presented for each individual pneumococcal conjugate serotype Opsonophagocytic Activity (OPA).
Time Frame: At 1 month after vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 411 | 408
Titers
  MOPA-1 | 67.6 [56.9 to 80.2] | 65.6 [55.2 to 77.9]
  MOPA-3 | 105.0 [92.2 to 119.5] | 108.9 [95.7 to 124.1]
  MOPA-4: number analyzed (Participants) | 409 | 408
  MOPA-4 | 1264.1 [1089.9 to 1466.2] | 1117.2 [963.1 to 1296.1]
  MOPA-5 | 152.6 [129.1 to 180.3] | 159.8 [135.1 to 188.9]
  MOPA-6B: number analyzed (Participants) | 409 | 408
  MOPA-6B | 1536.8 [1307.9 to 1805.7] | 1666.6 [1418.0 to 1958.6]
  MOPA-7F: number analyzed (Participants) | 409 | 407
  MOPA-7F | 2491.3 [2179.8 to 2847.5] | 2324.7 [2033.3 to 2657.9]
  MOPA-9V: number analyzed (Participants) | 410 | 406
  MOPA-9V | 1911.8 [1651.6 to 2212.9] | 1970.3 [1700.9 to 2282.3]
  MOPA-14: number analyzed (Participants) | 411 | 407
  MOPA-14 | 2610.1 [2281.6 to 2986.0] | 2678.1 [2339.4 to 3065.8]
  MOPA-18C: number analyzed (Participants) | 411 | 405
  MOPA-18C | 1040.9 [902.7 to 1200.4] | 1099.8 [952.8 to 1269.6]
  MOPA-19A: number analyzed (Participants) | 406 | 406
  MOPA-19A | 1558.6 [1361.8 to 1783.8] | 1350.5 [1180.0 to 1545.7]
  MOPA-19F: number analyzed (Participants) | 409 | 407
  MOPA-19F | 938.2 [814.6 to 1080.7] | 914.1 [793.4 to 1053.3]
  MOPA-23F: number analyzed (Participants) | 410 | 405
  MOPA-23F | 372.8 [316.0 to 439.8] | 419.1 [354.9 to 494.9]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of GMTs between groups (Control group and Co-Ad group) for MOPA-1; Test type: Non-Inferiority — Non Inferiority criterion used: Upper Limit (UL) of the 95% CI for each individual pneumococcal conjugate serotype Opsonophagocytic Assay (OPA) GMT ratio of the Control group over the Co-Ad group had to be below 2; ANCOVA; Ancova model: adjustment for baseline titre - pooled variance; Adjusted GMT = 1.03, 95% CI 2-sided [0.81 to 1.31] — Adjusted GMT ratio (Control group / Co-Ad group)
Statistical Analysis 2: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of GMTs between groups (Control group and Co-Ad group) for MOPA-3; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titre - pooled variance; Adjusted GMT = 0.96, 95% CI 2-sided [0.8 to 1.16] — Adjusted GMT ratio (Control group / Co-Ad group)
Statistical Analysis 3: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of GMTs between groups (Control group and Co-Ad group) for MOPA-4; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titre - pooled variance; Adjusted GMT = 1.13, 95% CI 2-sided [0.92 to 1.4] — Adjusted GMT ratio (Control group / Co-Ad group)
Statistical Analysis 4: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of GMTs between groups (Control group and Co-Ad group) for MOPA-5; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titre - pooled variance; Adjusted GMT = 0.96, 95% CI 2-sided [0.75 to 1.21] — Adjusted GMT ratio (Control group / Co-Ad group)
Statistical Analysis 5: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of GMTs between groups (Control group and Co-Ad group) for MOPA-6B; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titre - pooled variance; Adjusted GMT = 0.92, 95% CI 2-sided [0.73 to 1.16] — Adjusted GMT ratio (Control group / Co-Ad group)
Statistical Analysis 6: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of GMTs between groups (Control group and Co-Ad group) for MOPA-7F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titre - pooled variance; Adjusted GMT = 1.07, 95% CI 2-sided [0.89 to 1.29] — Adjusted GMT ratio (Control group / Co-Ad group)
Statistical Analysis 7: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of GMTs between groups (Control group and Co-Ad group) for MOPA-9V; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titre - pooled variance; Adjusted GMT = 0.97, 95% CI 2-sided [0.79 to 1.19] — Adjusted GMT ratio (Control group / Co-Ad group)
Statistical Analysis 8: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of GMTs between groups (Control group and Co-Ad group) for MOPA-14; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titre - pooled variance; Adjusted GMT = 0.97, 95% CI 2-sided [0.81 to 1.18] — Adjusted GMT ratio (Control group / Co-Ad group)
Statistical Analysis 9: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of GMTs between groups (Control group and Co-Ad group) for MOPA-18C; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titre - pooled variance; Adjusted GMT = 0.95, 95% CI 2-sided [0.77 to 1.16] — Adjusted GMT ratio (Control group / Co-Ad group)
Statistical Analysis 10: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of GMTs between groups (Control group and Co-Ad group) for MOPA-19A; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titre - pooled variance; Adjusted GMT = 1.15, 95% CI 2-sided [0.95 to 1.4] — Adjusted GMT ratio (Control group / Co-Ad group)
Statistical Analysis 11: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of GMTs between groups (Control group and Co-Ad group) for MOPA-19F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titre - pooled variance; Adjusted GMT = 1.03, 95% CI 2-sided [0.84 to 1.25] — Adjusted GMT ratio (Control group / Co-Ad group)
Statistical Analysis 12: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of GMTs between groups (Control group and Co-Ad group) for MOPA-23F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; ANCOVA; Ancova model: adjustment for baseline titre - pooled variance; Adjusted GMT = 0.89, 95% CI 2-sided [0.7 to 1.12] — Adjusted GMT ratio (Control group / Co-Ad group)

5. Primary Outcome: Adjusted GMCs Between Groups
Description: The Adjusted ratios of GMCs between groups (Control group and Co-Ad group) was presented for anti-gE antibody ELISA concentrations
Time Frame: At 1 month after last vaccine dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 401 | 402
mIU/mL | 49569.0 [46641.4 to 52680.4] | 50474.5 [47497.4 to 53638.2]
Statistical Analysis 1: Comparison: Co-Ad Group vs Control Group; Adjusted ratios of GMCs between groups (Control group and Co-Ad group) for anti-gE antibody ELISA concentrations; Test type: Non-Inferiority — Non Inferiority criterion used: UL of the 95% CI for the anti-gE antibodies GMC ratio between the Control group and the Co-Ad group had to be below 1.5; ANCOVA; Ancova model: adjustment for baseline concentration and age - pooled variance; Adjusted GMC = 1.02, 95% CI 2-sided [0.93 to 1.11] — Adjusted ratios of GMCs between groups (Control group and Co-Ad group)

6. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms, by Dose
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site. The Co-Ad Group received only 2 vaccine doses.
Time Frame: Within 7 days (Days 0 - 6) after each vaccination
Population: The analyses were performed on the Total Vaccinated cohort, which included all subjects with at least one administered vaccine and with the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 429 | 431
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 428 | 431
  Any Pain, Dose 1 | 344 | 169
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 428 | 431
  Grade 3 Pain, Dose 1 | 46 | 5
  Any Redness, Dose 1: number analyzed (Participants) | 428 | 431
  Any Redness, Dose 1 | 182 | 31
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 428 | 431
  Grade 3 Redness, Dose 1 | 15 | 2
  Any Swelling, Dose 1: number analyzed (Participants) | 428 | 431
  Any Swelling, Dose 1 | 99 | 21
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 428 | 431
  Grade 3 Swelling, Dose 1 | 4 | 1
  Any Pain, Dose 2: number analyzed (Participants) | 416 | 422
  Any Pain, Dose 2 | 298 | 290
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 416 | 422
  Grade 3 Pain, Dose 2 | 35 | 28
  Any Redness, Dose 2: number analyzed (Participants) | 416 | 422
  Any Redness, Dose 2 | 146 | 129
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 416 | 422
  Grade 3 Redness, Dose 2 | 15 | 4
  Any Swelling, Dose 2: number analyzed (Participants) | 416 | 422
  Any Swelling, Dose 2 | 79 | 67
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 416 | 422
  Grade 3 Swelling, Dose 2 | 4 | 2
  Any Pain, Dose 3: number analyzed (Participants) | 0 | 419
  Any Pain, Dose 3 | 0 | 293
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 0 | 419
  Grade 3 Pain, Dose 3 | 0 | 32
  Any Redness, Dose 3: number analyzed (Participants) | 0 | 419
  Any Redness, Dose 3 | 0 | 136
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 0 | 419
  Grade 3 Redness, Dose 3 | 0 | 8
  Any Swelling, Dose 3: number analyzed (Participants) | 0 | 419
  Any Swelling, Dose 3 | 0 | 74
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 0 | 419
  Grade 3 Swelling, Dose 3 | 0 | 3
  Any Pain, Across Doses | 372 | 357
  Grade 3 Pain, Across Doses | 68 | 49
  Any Redness, Across Doses | 233 | 194
  Grade 3 Redness, Across Doses | 27 | 12
  Any Swelling, Across Doses | 137 | 115
  Grade 3 Swelling, Across Doses | 7 | 6

7. Secondary Outcome: Number of Subjects With Solicited Local Symptoms, Across Doses, by Vaccine
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: Within 7 days (Days 0 - 6) after vaccination
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 429 | 431
Participants
  Any Pain, GSK1437173A, Across Doses: number analyzed (Participants) | 429 | 426
  Any Pain, GSK1437173A, Across Doses | 369 | 343
  Any Pain, Pneumovax 23, Across Doses: number analyzed (Participants) | 428 | 431
  Any Pain, Pneumovax 23, Across Doses | 223 | 169
  Any Redness, GSK1437173A, Across Doses | 223 | 186
  Any Redness, Pneumovax 23, Across Doses: number analyzed (Participants) | 428 | 431
  Any Redness, Pneumovax 23, Across Doses | 69 | 31
  Any Swelling, GSK1437173A, Across Doses: number analyzed (Participants) | 429 | 426
  Any Swelling, GSK1437173A, Across Doses | 129 | 108
  Any Swelling, Pneumovax 23, Across Doses: number analyzed (Participants) | 428 | 431
  Any Swelling, Pneumovax 23, Across Doses | 36 | 21

8. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], headache, myalgia, shivering and sweating. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: This analysis was performed on the Total Vaccinated cohort, including subjects with at least one vaccine dose administered, only on those subjects with completed symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 429 | 431
Participants
  Any Fatigue, Dose 1: number analyzed (Participants) | 427 | 430
  Any Fatigue, Dose 1 | 194 | 87
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 427 | 430
  Grade 3 Fatigue, Dose 1 | 27 | 3
  Related Fatigue, Dose 1: number analyzed (Participants) | 427 | 430
  Related Fatigue, Dose 1 | 175 | 81
  Any Gastrointestinal symptoms, Dose 1: number analyzed (Participants) | 427 | 430
  Any Gastrointestinal symptoms, Dose 1 | 76 | 31
  Grade 3 Gastrointestinal symptoms, Dose 1: number analyzed (Participants) | 427 | 430
  Grade 3 Gastrointestinal symptoms, Dose 1 | 6 | 1
  Related Gastrointestinal symptoms, Dose 1: number analyzed (Participants) | 427 | 430
  Related Gastrointestinal symptoms, Dose 1 | 67 | 28
  Any Headache, Dose 1: number analyzed (Participants) | 427 | 430
  Any Headache, Dose 1 | 156 | 72
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 427 | 430
  Grade 3 Headache, Dose 1 | 15 | 3
  Related Headache, Dose 1: number analyzed (Participants) | 427 | 430
  Related Headache, Dose 1 | 141 | 64
  Any Myalgia, Dose 1: number analyzed (Participants) | 427 | 430
  Any Myalgia, Dose 1 | 187 | 87
  Grade 3 Myalgia, Dose 1: number analyzed (Participants) | 427 | 430
  Grade 3 Myalgia, Dose 1 | 29 | 5
  Related Myalgia, Dose 1: number analyzed (Participants) | 427 | 430
  Related Myalgia, Dose 1 | 177 | 82
  Any Shivering, Dose 1: number analyzed (Participants) | 427 | 430
  Any Shivering, Dose 1 | 91 | 27
  Grade 3 Shivering, Dose 1: number analyzed (Participants) | 427 | 430
  Grade 3 Shivering, Dose 1 | 12 | 1
  Related Shivering, Dose 1: number analyzed (Participants) | 427 | 430
  Related Shivering, Dose 1 | 86 | 26
  Any Temperature, Dose 1: number analyzed (Participants) | 427 | 430
  Any Temperature, Dose 1 | 69 | 12
  Grade 3 Temperature, Dose 1: number analyzed (Participants) | 427 | 430
  Grade 3 Temperature, Dose 1 | 1 | 1
  Related Temperature, Dose 1: number analyzed (Participants) | 427 | 430
  Related Temperature, Dose 1 | 67 | 11
  Any Fatigue, Dose 2: number analyzed (Participants) | 415 | 421
  Any Fatigue, Dose 2 | 191 | 124
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 415 | 421
  Grade 3 Fatigue, Dose 2 | 29 | 11
  Related Fatigue, Dose 2: number analyzed (Participants) | 415 | 421
  Related Fatigue, Dose 2 | 174 | 109
  Any Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 415 | 421
  Any Gastrointestinal symptoms, Dose 2 | 61 | 38
  Grade 3 Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 415 | 421
  Grade 3 Gastrointestinal symptoms, Dose 2 | 6 | 4
  Related Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 415 | 421
  Related Gastrointestinal symptoms, Dose 2 | 52 | 29
  Any Headache, Dose 2: number analyzed (Participants) | 415 | 421
  Any Headache, Dose 2 | 141 | 104
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 415 | 421
  Grade 3 Headache, Dose 2 | 19 | 9
  Related Headache, Dose 2: number analyzed (Participants) | 415 | 421
  Related Headache, Dose 2 | 124 | 85
  Any Myalgia, Dose 2: number analyzed (Participants) | 415 | 421
  Any Myalgia, Dose 2 | 182 | 124
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 415 | 421
  Grade 3 Myalgia, Dose 2 | 25 | 11
  Related Myalgia, Dose 2: number analyzed (Participants) | 415 | 421
  Related Myalgia, Dose 2 | 171 | 119
  Any Shivering, Dose 2: number analyzed (Participants) | 415 | 421
  Any Shivering, Dose 2 | 83 | 30
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 415 | 421
  Grade 3 Shivering, Dose 2 | 14 | 3
  Related Shivering, Dose 2: number analyzed (Participants) | 415 | 421
  Related Shivering, Dose 2 | 78 | 25
  Any Temperature, Dose 2: number analyzed (Participants) | 415 | 421
  Any Temperature, Dose 2 | 67 | 30
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 415 | 421
  Grade 3 Temperature, Dose 2 | 0 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 415 | 421
  Related Temperature, Dose 2 | 63 | 26
  Any Fatigue, Dose 3: number analyzed (Participants) | 0 | 419
  Any Fatigue, Dose 3 | 0 | 174
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 0 | 419
  Grade 3 Fatigue, Dose 3 | 0 | 22
  Related Fatigue, Dose 3: number analyzed (Participants) | 0 | 419
  Related Fatigue, Dose 3 | 0 | 166
  Any Gastrointestinal symptoms, Dose 3: number analyzed (Participants) | 0 | 419
  Any Gastrointestinal symptoms, Dose 3 | 0 | 47
  Grade 3 Gastrointestinal symptoms, Dose 3: number analyzed (Participants) | 0 | 419
  Grade 3 Gastrointestinal symptoms, Dose 3 | 0 | 3
  Related Gastrointestinal symptoms, Dose 3: number analyzed (Participants) | 0 | 419
  Related Gastrointestinal symptoms, Dose 3 | 0 | 46
  Any Headache, Dose 3: number analyzed (Participants) | 0 | 419
  Any Headache, Dose 3 | 0 | 144
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 0 | 419
  Grade 3 Headache, Dose 3 | 0 | 13
  Related Headache, Dose 3: number analyzed (Participants) | 0 | 419
  Related Headache, Dose 3 | 0 | 135
  Any Myalgia, Dose 3: number analyzed (Participants) | 0 | 419
  Any Myalgia, Dose 3 | 0 | 162
  Grade 3 Myalgia, Dose 3: number analyzed (Participants) | 0 | 419
  Grade 3 Myalgia, Dose 3 | 0 | 26
  Related Myalgia, Dose 3: number analyzed (Participants) | 0 | 419
  Related Myalgia, Dose 3 | 0 | 157
  Any Shivering, Dose 3: number analyzed (Participants) | 0 | 419
  Any Shivering, Dose 3 | 0 | 72
  Grade 3 Shivering, Dose 3: number analyzed (Participants) | 0 | 419
  Grade 3 Shivering, Dose 3 | 0 | 11
  Related Shivering, Dose 3: number analyzed (Participants) | 0 | 419
  Related Shivering, Dose 3 | 0 | 69
  Any Temperature, Dose 3: number analyzed (Participants) | 0 | 419
  Any Temperature, Dose 3 | 0 | 67
  Grade 3 Temperature, Dose 3: number analyzed (Participants) | 0 | 419
  Grade 3 Temperature, Dose 3 | 0 | 2
  Related Temperature, Dose 3: number analyzed (Participants) | 0 | 419
  Related Temperature, Dose 3 | 0 | 66
  Any Fatigue, Across doses | 253 | 228
  Grade 3 Fatigue, Across doses | 47 | 31
  Related Fatigue, Across doses | 236 | 216
  Any Gastrointestinal symptoms, Across doses | 114 | 84
  Grade 3 Gastrointestinal symptoms, Across doses | 12 | 7
  Related Gastrointestinal symptoms, Across doses | 100 | 77
  Any Headache, Across doses | 209 | 208
  Grade 3 Headache, Across doses | 29 | 24
  Related Headache, Across doses | 195 | 193
  Any Myalgia, Across doses | 257 | 225
  Grade 3 Myalgia, Across doses | 46 | 37
  Related Myalgia, Across doses | 245 | 218
  Any Shivering, Across doses | 137 | 99
  Grade 3 Shivering, Across doses | 25 | 15
  Related Shivering, Across doses | 131 | 95
  Any Temperature, Across doses | 112 | 96
  Grade 3 Temperature, Across doses | 1 | 3
  Related Temperature, Across doses | 108 | 91

9. Secondary Outcome: Number of Days With Any Solicited Local and General Symptoms
Description: The Co-Ad Group received only 2 vaccine doses, hence the number of participants for the Dose 3 categories in this group is 0.
Time Frame: Within 7 days (Days 0 - 6) after each vaccination
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Co-Ad Group: Subjects received one dose of the GSK1437173A study vaccine and one dose of the Pneumovax™ 23 vaccine at Day 0 and a second dose of GSK1437173A study vaccine at Month 2. GSK1437173A vaccine was administered intramuscularly, in the deltoid region of the non-dominant arm. Pneumovax™ 23 was administered intramuscularly, in the deltoid region of the dominant arm .
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 344 | 293
days
  Any Pain, Dose 1: number analyzed (Participants) | 344 | 169
  Any Pain, Dose 1 | 3 [2 to 4] | 2 [1 to 3]
  Any Pain, Dose 2: number analyzed (Participants) | 298 | 290
  Any Pain, Dose 2 | 3 [2 to 4] | 3 [2 to 4]
  Any Pain, Dose 3: number analyzed (Participants) | 0 | 293
  Any Pain, Dose 3 |  | 3 [2 to 4]
  Any Redness, Dose 1: number analyzed (Participants) | 182 | 31
  Any Redness, Dose 1 | 3 [2 to 5] | 2 [1 to 3]
  Any Redness, Dose 2: number analyzed (Participants) | 146 | 129
  Any Redness, Dose 2 | 3 [2 to 4] | 3 [2 to 5]
  Any Redness, Dose 3: number analyzed (Participants) | 0 | 136
  Any Redness, Dose 3 |  | 3 [2 to 4]
  Any Swelling, Dose 1: number analyzed (Participants) | 99 | 21
  Any Swelling, Dose 1 | 3 [2 to 5] | 2 [1 to 3]
  Any Swelling, Dose 2: number analyzed (Participants) | 79 | 67
  Any Swelling, Dose 2 | 3 [2 to 4] | 4 [2 to 5]
  Any Swelling, Dose 3: number analyzed (Participants) | 0 | 74
  Any Swelling, Dose 3 |  | 3 [2 to 5]
  Any Fatigue, Dose 1: number analyzed (Participants) | 194 | 87
  Any Fatigue, Dose 1 | 2 [1 to 4] | 2 [1 to 4]
  Any Fatigue, Dose 2: number analyzed (Participants) | 191 | 124
  Any Fatigue, Dose 2 | 2 [1 to 3] | 2 [1 to 3]
  Any Fatigue, Dose 3: number analyzed (Participants) | 0 | 174
  Any Fatigue, Dose 3 |  | 2 [1 to 3]
  Any Gastrointestinal, Dose 1: number analyzed (Participants) | 76 | 31
  Any Gastrointestinal, Dose 1 | 2 [1 to 2.5] | 2 [1 to 3]
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 61 | 38
  Any Gastrointestinal, Dose 2 | 2 [1 to 3] | 2 [1 to 3]
  Any Gastrointestinal, Dose 3: number analyzed (Participants) | 0 | 47
  Any Gastrointestinal, Dose 3 |  | 2 [1 to 2]
  Any Headache, Dose 1: number analyzed (Participants) | 156 | 72
  Any Headache, Dose 1 | 2 [1 to 3] | 2 [1 to 2]
  Any Headache, Dose 2: number analyzed (Participants) | 141 | 104
  Any Headache, Dose 2 | 2 [1 to 3] | 2 [1 to 2.5]
  Any Headache, Dose 3: number analyzed (Participants) | 0 | 144
  Any Headache, Dose 3 |  | 2 [1 to 2]
  Any Myalgia, Dose 1: number analyzed (Participants) | 187 | 87
  Any Myalgia, Dose 1 | 2 [2 to 4] | 2 [1 to 3]
  Any Myalgia, Dose 2: number analyzed (Participants) | 182 | 124
  Any Myalgia, Dose 2 | 2 [1 to 3] | 2 [1 to 3.5]
  Any Myalgia, Dose 3: number analyzed (Participants) | 0 | 162
  Any Myalgia, Dose 3 |  | 2 [2 to 3]
  Any Shivering, Dose 1: number analyzed (Participants) | 91 | 27
  Any Shivering, Dose 1 | 1 [1 to 2] | 2 [1 to 2]
  Any Shivering, Dose 2: number analyzed (Participants) | 83 | 30
  Any Shivering, Dose 2 | 1 [1 to 2] | 1 [1 to 2]
  Any Shivering, Dose 3: number analyzed (Participants) | 0 | 72
  Any Shivering, Dose 3 |  | 1 [1 to 2]
  Any Temperature (Oral), Dose 1: number analyzed (Participants) | 69 | 12
  Any Temperature (Oral), Dose 1 | 1 [1 to 2] | 1 [1 to 2]
  Any Temperature (Oral), Dose 2: number analyzed (Participants) | 67 | 30
  Any Temperature (Oral), Dose 2 | 1 [1 to 2] | 1 [1 to 2]
  Any Temperature (Oral), Dose 3: number analyzed (Participants) | 0 | 67
  Any Temperature (Oral), Dose 3 |  | 1 [1 to 2]

10. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: From the first dose up to 30 days post last vaccination period
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 432 | 433
Participants
  Subjects with any AE(s) | 132 | 140
  Subjects with grade 3 AE(s) | 16 | 28
  Subjects with related AE(s) | 34 | 28

11. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) [From the First Dose up to 30 Days Post Last Vaccination Period]
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From the first dose up to 30 days post last vaccination period
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 432 | 433
Participants
  Subjects with any SAE(s) | 7 | 9
  Fatal SAEs | 0 | 0

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) [From 30 Days Post Last Vaccination up to Study End]
Description: as for outcome 11
Time Frame: From 30 days post last vaccination up to study end
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 432 | 433
Participants
  Subjects with any SAE(s) | 10 | 10
  Fatal SAE(s) | 2 | 2
  Related SAE(s) | 2 | 2

13. Secondary Outcome: Number of Subjects With Potential Immune Mediated Diseases (pIMDs) [From First Vaccination up to 30 Days Post Last Vaccination]
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From first vaccination up to 30 days post last vaccination (Month 0 - Month 3 for the Co-Ad Group & Month 0 - Month 5 for the Control Group)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 432 | 433
Participants
  Any pIMDs | 0 | 1
  Related pIMDs | 0 | 0

14. Secondary Outcome: Number of Subjects With Potential Immune Mediated Diseases (pIMDs) [During the Period Starting After 30 Days Post Last Vaccination up to Study End]
Description: as for outcome 13
Time Frame: During the period starting after 30 days post last vaccination up to study end (Month 3 - Month 14 for the Co-Ad Group & Month 5 - Month 16 for the Control Group)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Co-Ad Group | Control Group
Number analyzed (Participants) | 432 | 433
Participants | 1 | 0

ADVERSE EVENTS:
Arm/Group | Co-Ad Group | Control Group
All-Cause Mortality (participants affected / at risk) | 2/432 | 5/433
Serious Adverse Events (participants affected / at risk) | 17/432 | 19/433
Other Adverse Events (participants affected / at risk) | 400/432 | 393/433
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Ad Group (N=432) | Control Group (N=433)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral artery dissection (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Ad Group (N=432) | Control Group (N=433)
Gastrointestinal disorder (Gastrointestinal disorders) | 114 (137) | 84 (116)
Chills (Gastrointestinal disorders) | 137 (176) | 99 (130)
Fatigue (General disorders) | 253 (385) | 228 (385)
Pain (General disorders) | 372 (642) | 357 (754)
Pyrexia (General disorders) | 112 (138) | 97 (110)
Swelling (General disorders) | 137 (178) | 115 (162)
Myalgia (Musculoskeletal and connective tissue disorders) | 257 (370) | 227 (376)
Headache (Nervous system disorders) | 210 (306) | 209 (331)
Erythema (General disorders) | 234 (330) | 194 (297)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.